CLINICAL TRIAL: NCT06575166
Title: The Impact of Abdominal Wall Reconstruction on Abdominal Wall Tension and Intra-Abdominal Pressure
Status: Terminated | Type: Observational
Why Stopped: Interoperability issue between necessary devices.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Benjamin T. Miller, Principal Investigator, The Cleveland Clinic
Other Study IDs: 24-655
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2024-08

CONDITIONS: Ventral Hernia; Incisional Hernia; Parastomal Hernia
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Abdominal wall tension — Abdominal wall tension measurement All patients will have the tension of their abdominal wall measured during surgery using a tension scale or "tensiometer."
  Other Names: Tensiometry
Device: Intra-abdominal pressure — Intra-abdominal pressure All patients will have their intra-abdominal pressure continuously monitored using Sentinel's FDA approved TraumaGuard catheter, a pressure-sensing urinary catheter.
  Other Names: IAP

SUMMARY:
This is a prospective cohort study. Patients have an incisional or parastomal hernia with >20 cm fascial defect on pre-operative imaging who will undergo an anticipated open bilateral transversus abdominis release with retromuscular synthetic mesh will have their abdominal wall tension measured using a tension scale and their intra-abdominal pressure measured using a urinary catheter containing pressure sensors. The investigators aim to quantify the changes, as well as explore and describe the physiologic shifts that may be associated with these changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Incisional or parastomal hernia with >20 cm fascial defect on pre-operative imaging
* Anticipated open bilateral transversus abdominis release with retro-muscular synthetic mesh placement

Exclusion Criteria:

* Pregnant patients
* Require a Legally Authorized Representative (LAR) to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with an incisional or parastomal hernia with a >20 cm fascial defect on pre-operative imaging who undergo an anticipated open bilateral transversus abdominis release with retro-muscular synthetic mesh placement will be included. The investigators anticipate that patients with very large defects will experience the greatest changes in abdominal wall tension and intra-abdominal pressure.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Correlation between intra-abdominal pressure (mmHg) and rate of post-operative complications | 1 year
  Intra-abdominal pressure measured in mmHg using TraumaGuard catheter Post-operative complications measured in proportion of events

SECONDARY OUTCOMES:
Correlation between intra-abdominal pressure (mmHg) to abdominal wall tension (lbs) | 1 year
  Intra-abdominal pressure measured in mmHg using TraumaGuard catheter Abdominal wall tension measured using tensiometer in pounds (lbs)
Correlation between abdominal wall tension (lbs) and intra-abdominal pressure (mmHg) to hernia defect size (cm) | 1 year
  Intra-abdominal pressure measured in mmHg using TraumaGuard catheter Abdominal wall tension measured using tensiometer in pounds (lbs) Hernia defect size (length and width in cm)
Correlation between abdominal wall tension (lbs) and intra-abdominal pressure (mmHg) to airway pressure (cmH2O) | 1 year
  Intra-abdominal pressure using TraumaGuard catheter in mmHg Abdominal wall tension measured using tensiometer in pounds Airway pressure measured on mechanical ventilator in cmH2O
Temporal changes in renal function (serum Creatinine) | 1 year
  Creatinine reported on routine laboratory blood work (comprehensive metabolic panel) measured over time

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Miller, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No